CLINICAL TRIAL: NCT00942799
Title: A Phase I, Open-Label, Multicenter, Dose Escalation Study to Assess the Safety and Tolerability of Genz-644282 in Patients With Advanced Malignant Solid Tumors
Brief Title: Dose Escalation Study to Assess the Safety and Tolerability of Genz-644282 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZ28200108
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Solid Tumors
Keywords: Genz-644282; Topoisomerase I inhibitors; Top1; solid tumors; dose-escalation; pharmacokinetic (PK); MTD (Maximum Tolerated Dose); oncology; cancer
MeSH Terms: conditions — Metatropic dwarfism; Neoplasms | interventions — Genz-644282

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Drug: Genz-644282 (28-day dosing schedule) (Experimental): Genz-644282 (Each cohort will be based on dose-escalation)
  Interventions: Drug: Genz-644282 (28-day dosing schedule)
- Study Drug: Genz-644282 (21-day dosing schedule) (Experimental): Genz-644282 (Each cohort will be based on dose-escalation)
  Interventions: Drug: Genz-644282 (21-day dosing schedule)

INTERVENTIONS:
Drug: Genz-644282 (28-day dosing schedule) — Genz-644282 will be administered as a 60-minute IV infusion. The initial dose of Genz-644282 will be 0.5 mg/m2 and will be administered once weekly for 3 consecutive weeks on Day 1, Day 8, and Day 15 of the 28 day cycle. Each 28-day period will represent one treatment cycle. Study drug will continue to be given until disease progression or unacceptable toxicity is observed.
  Arms: Study Drug: Genz-644282 (28-day dosing schedule)
Drug: Genz-644282 (21-day dosing schedule) — The starting dose of Genz-644282 for the 21-day schedule will be prescriptive and will be based on review of available safety data from the 28-day dosing schedule by the Investigator and Sponsor. Patients will receive Genz-644282 once-weekly for 2 consecutive weeks on Day 1 and Day 8 of a 21 day cycle. Each 21-day period will represent 1 treatment cycle. Patients enrolled in subsequent cohorts will receive higher doses until the MTD is established.
  Arms: Study Drug: Genz-644282 (21-day dosing schedule)

SUMMARY:
This is a Phase I, open-label, multicenter, dose-escalation study designed to assess the safety and tolerability of Genz-644282, administered as an intravenous (IV) infusion, to patients with advanced malignant solid tumors. Each 28 day cycle of treatment will consist of 3 consecutive weeks of treatment every 28 days(i.e., treatment will be administered on Days 1, 8, and 15 every 28 days). Each 21 day cycle of treatment will consist of 2 consecutive weeks of treatment every 21 days(i.e., treatment will be administered on Days 1 and 8 every 21 days). Treatment with Genz-644282 will continue until disease progression or unacceptable toxicity is observed. Approximately 110 patients will be enrolled in this study. Patients will be enrolled in escalating dose cohorts until the Maximum Tolerated Doses (MTDs) for the 2 dosing schedules are established. To further evaluate safety, approximately 40 additional patients with advanced malignant solid tumors will be enrolled and treated at the MTDs (20 for each dosing schedule) during an expansion phase.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multicenter, dose-escalation study designed to assess the safety and tolerability of Genz-644282, administered as an IV infusion, to patients with advanced malignant solid tumors. Drug will be administered as a 60-minute IV infusion on days 1, 8, and 15 of the 28 day treatment cycle, or on days 1 and 8 of the 21 day treatment cycle.

Treatment with Genz-644282 will continue until disease progression or unacceptable toxicity is observed. Patients will be enrolled in escalating dose cohorts until the Maximum Tolerated Doses (MTDs) are established.

Safety will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients enrolled in dose-escalation phase: Histologically or cytologically confirmed advanced malignant solid tumor for which no standard therapeutic option exists.
* For the disease indications evaluated in the expansion phase, the following criteria must be met:

  1. Have one of the following histologically or cytologically confirmed advanced malignant solid tumors for which no standard therapeutic option exists:

     * Colorectal cancer (prior systemic regimen must have included ≥1 of the following: fluoropyrimidine or oxaliplatin);
     * Squamous Non-small cell lung cancer or small cell lung cancer (prior systemic regimen must have included ≥1 of the following: cis-platinum or carbo platinum);
     * Pancreatic cancer (prior systemic regimen must have included gemcitabine);
     * Breast cancer (prior systemic regimen must have included ≥1 of the following: taxane, anthracycline, or fluoropyrimidine)
  2. Received no more than 4 prior systemic therapy regimens for their malignancy
  3. Experienced progression or intolerance to their immediate prior systemic therapy regimen.
* Evaluable or measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 12 weeks.
* Adequate organ and hematologic function.
* Prior chemotherapy, major surgery, or irradiation must have been completed at least 3 weeks prior to starting treatment with study drug, with the exception of mitomycin-C or nitrosoureas, which should be completed at least 6 weeks prior. Additionally, patients must have recovered to ≤ Grade 1 toxicities incurred as a result of the previous therapy, with the exception of nail dystrophy, alopecia, or local radiation therapy induced adverse events (e.g., impotence or incontinence). A patient who has received radiation to < 5% of their total bone marrow volume and who has had 2 weeks of rest may be considered for study entry after discussion with the Sponsor
* Hormone treatment must have been completed > 2 weeks prior to receiving study drug.
* Prostate cancer patients who are chemically castrated with hormonal therapy (e.g., luteinizing hormone-releasing hormone agonists) will be allowed to enter the study. However, doses and schedules of such treatments must be maintained throughout the trial and all major toxicities must have resolved to ≤ Grade 1 prior to study entry.
* Concomitant stable treatment with bisphosphonates is allowed, unless dose requires readjustments or discontinuation.
* Ability to comply with study procedures and follow-up examinations.
* Male and female patients must agree to use an effective barrier means of birth control (i.e., latex condom, diaphragm, cervical cap, etc.) throughout the entire duration of the study and for at least 3 months after last dose of study drug.
* Male patients must agree to not donate sperm throughout the study and for at least 3 months following the last dose of study drug.

Exclusion Criteria:

* Received previous treatment with or have a known hypersensitivity to Genz-644282 or to any of its components.
* Received radiotherapy to the only site of measurable disease, unless the tumor at this site continues to increase in size after the patient has completed radiotherapy treatment.
* Used any investigational agent, other than anti-cancer chemotherapy, during the 4 weeks prior to the first dose of Genz-644282.
* Have psychiatric disorder(s) that would interfere with consent, study participation, or follow up (with the possible exception of incompetence as defined by New Jersey for the purposes of participation in clinical trials in the state of New Jersey).
* Have uncontrolled congestive heart failure or angina, a history of myocardial infarction within 6 months prior to study enrollment, or a cardiac functional capacity Class III or IV, as defined by the New York Heart Association Classification.
* Have a resting QT with Bazett's correction (QTcB) interval of > 460 msec, calculated as the average of at least 2 of the longest QT intervals measured on 12-lead recordings made prior to dosing with Genz-644282.
* Have a systemic fungal, bacterial, viral, or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement) despite appropriate antibiotics or other treatment.
* Have any other severe concurrent disease or a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo chemotherapy.
* A known diagnosis of human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS) or viral hepatitis B or C.
* Presence of ≥ Grade 2 peripheral neuropathy.
* Pregnant or lactating women, due to the unknown effects of Genz-644282 on the developing fetus or newborn infant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Doses for the 28-day and 21-day dosing schedules | 24 Months

SECONDARY OUTCOMES:
Determine the recommended Phase 2 doses for the 28-day and 21-day dosing schedules | 36 Months
Establish the pharmacokinetic (PK) profile through calculation of area under the curve of blood and urine concentrations. | 36 Months
Pharmacokinetics (PK) as measured by maximal observed concentration (Cmax) | 36 months
Pharmacokinetics (PK) as measured by time to maximal observed concentration (Tmax) | 36 months
Pharmacokinetics (PK) as measured by half-life (T1/2) | 36 months
Pharmacokinetics (PK) as measured by the amount and fraction of drug excreted in urine | 36 months
Assess evidence of antitumor activity | 36 months
Evaluate ongoing benefit as determined by the investigator and defined as an improvement in performance status | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (4):
- United States (4):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - Moffitt Cancer Center, Tampa, Florida
  - Wayne State University, Division of Hematology/Oncology, Karmanos Cancer Institute, Detroit, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey